CLINICAL TRIAL: NCT05136911
Title: South Asian Low-sodium Trial: A Pilot Randomized Controlled Trial
Brief Title: South Asian Low-sodium Trial
Acronym: SALT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment was stopped due to province-wide lockdown secondary to COVID-19. Blood pressure screenings were conducted in community centres and due to province wide lockdown, further screenings could not be continued.
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Salima Hemani, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 37070
Record Dates: First submitted 2021-10-15; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A pragmatic two-arm parallel 6-week randomized controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will be responsible for randomization and the outcome assessor (research assistant) will be blinded to group allocation. The research assistant will collect all outcome data at 6 weeks from the intervention and usual care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive the standard care in the form of HTN Canada Booklet, advice to see their health care provider, urgent care or walk-in clinic and the Salt Intervention (Salt Intervention Manual, five weekly online modules and five weekly telephone calls.
  Interventions: Behavioral: SALT-Intervention
- Usual Care Group (No Intervention): All participants in the usual care group will receive the standard care in the form of HTN Canada Booklet, advice to see their health care provider, urgent care of walk-in clinic.

INTERVENTIONS:
Behavioral: SALT-Intervention — Participants in the intervention group will have access to all standard care as provided to the usual care group participants. In addition, participants in the intervention group will receive the SALT-intervention developed by the principal investigator in the form of a SALT-intervention consist of the Salt Intervention manual, five online modules which include a virtual cooking demonstration and five ten-minute weekly telephone calls delivered by the principal investigator.These strategies aim to increase knowledge, enhance self-management abilities and provide social support.
  Arms: Intervention Group

SUMMARY:
The overall goal of this pilot study is to examine the feasibility and acceptability of a culturally-tailored low-sodium dietary intervention is South Asian Canadians with stage one HTN. Specific objectives are to determine the feasibility (recruitment, retention, engagement and acceptability) of this intervention. Secondary outcomes include the effect of low-sodium dietary intervention on knowledge, attitude and self-regulation behaviours. Exploratory outcomes include its effect of systolic, diastolic blood pressure and sodium intake. Information obtained from this pilot trial will inform design of a larger randomized controlled trial in reducing BP in South Asian Canadians.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality and morbidity worldwide. Hypertension (HTN) is an important risk factor for cardiovascular disease. According to HTN Canada guidelines, HTN is classified as pre-hypertension (systolic BP of 120-139 mmHg or diastolic BP of 80-89 mmHg), stage one HTN ( systolic BP 140-159 mmHg or diastolic BP 90-99 mmHg) and stage two HTN (greater than or equal to systolic BP of 160 mmHg or greater than or equal to diastolic BP of 100 mmHg) (2). Any increase in blood pressure above optimal confers independent risk of cardiovascular disease, stroke, congestive heart failure, end-stage renal disease, peripheral vascular disease, dementia, atrial fibrillation and retinopathy. South Asian individuals have significantly higher rates of morbidity and mortality from cardiovascular diseases. Hypertension is prevalent in South Asian Canadians with prevalence rate of 17%. Hypertension is a result of various factors, which include excessive alcohol consumption. lack of dietary potassium, physical inactivity, obesity and high dietary sodium intake. High dietary sodium consumption is an important contributor to HTN. and the rapid increase in dietary sodium is contributing to the current epidemic of HTN and cardiovascular disease. Sodium has a positive linear causal relationship to blood pressure based on epidemiological and experimental studies. Sodium intake greater than 2300mg/day has been associated with an increased risk of developing HTN. In addition to HTN, excess sodium intake is associated with higher risk of developing dementia, osteoporosis, stomach cancer, left ventricular hypertrophy and heart failure. The average sodium intake of Canadians is currently estimated at 2760mg/day, which is well above the recommended daily intake of 2300mg/day. South Asians consume significantly higher amounts of sodium with more than 95% of South Asians add salt to their cooking. Sodium intake in South Asians has been reported in different countries as; 3456 mg/day in Pakistan, 3548-3708 mg/day in India, 5863-10,000mg/day in Bangladesh. Although dietary patterns vary considerably in South Asians, addition of salt during food preparation and at the table are common practices across communities. The combination of traditional as well as a western diet results in an increased amount of sodium from conveniently available traditional meals, consumption of bread, pizza, pasta and other processed foods, high sodium spices and addition of salt during cooking.

Interventions aimed at reducing dietary sodium reduces blood pressure as well as cardiovascular morbidity and mortality. Despite the known benefits of sodium reduction interventions in reducing blood pressure in the Caucasian population, there is limited research available to provide evidence that sodium reduction is beneficial in reducing blood pressure in South Asian Canadians with stage one HTN.

The primary purpose of the South Asian Low-sodium Trial (SALT) is to assess feasibility (recruitment, retention, engagement and acceptability) of implementing a six-week low-sodium community-based dietary intervention in South Asian Canadians with stage one HTN. Secondary objectives include assessing knowledge & attitude and self-regulation behaviours. Exploratory objectives are to assess change in systolic BP, diastolic BP and sodium intake.

ELIGIBILITY:
Inclusion Criteria:

1. South Asian individuals (India, Pakistan, Srilanka, Bangladesh, Nepal and Bhutan) over the age of 18 years
2. Stage one HTN, systolic BP of 140-159 mmHg or diastolic BP of 90-99 mmHg at baseline and not on anti-hypertensive medications
3. Consuming a daily sodium intake of >2000 mg/24 hours as determined at baseline by an online Salt Calculator,
4. Able to read, understand and write English
5. Access to computer with internet capabilities and a telephone

Exclusion Criteria:

1. Use of anti-hypertensive medications
2. Use of herbal or over-the counter medications to control BP
3. Use of insulin or oral hypoglycemic agents
4. Have an active cancer diagnosis or on treatment during the past three months due to interference between diet and cancer treatment
5. Have special dietary requirements and unable to consume a self-selected diet
6. Are pregnant, breastfeeding or anticipate pregnancy prior to the end of the study
7. Individuals who plan to leave the area prior to the anticipated end of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Recruitment | End of study-6 weeks
  Number of eligible participants agreeing to participate compared to total eligible participants
Retention | Through study completion-6 weeks
  Number of participants who complete follow-up assessment at 6-weeks.
Intervention Engagement with the SALT Intervention Manual | Through study completion, 6-weeks
  Number of participants in the intervention group who read the manual in its entirety
Intervention Engagement with five weekly online modules | Through study completion, 6-weeks
  Number of participants in the intervention group who complete the five weekly online modules
Intervention Engagement with five weekly goal-setting worksheets | Through study completion, 6-weeks
  Number of participants in the intervention group who complete the five goal-setting worksheets
Intervention Engagement with five weekly telephone calls | Through study completion, 6-weeks
  Number of participants in the intervention group who complete the five weekly telephone calls
Intervention Acceptability Questionnaire | Through study completion, 6-weeks
  Intervention Acceptability (Likert scale): Minimum Score: 0 and Maximum Score: 40, Higher score indicate higher acceptability
Intervention Acceptability-1 | Through study completion, 6-weeks
  Ease of reading SALT-Intervention Manual
Intervention Acceptability-2 | Through study completion, 6-weeks
  Ease of using goal-setting worksheets
Intervention Acceptability-3 | Through study completion, 6-weeks
  Ease of using online modules
Intervention Acceptability-4 | Through study completion, 6-weeks
  Ease of viewing cooking demonstration
Intervention Acceptability-6 | Through study completion, 6-weeks
  Ease of attending weekly telephone calls
Intervention Acceptability-7 | Through study completion, 6-weeks
  Encouragement to reduce sodium
Intervention Acceptability-8 | Through study completion, 6-weeks
  Satisfaction with time to complete study components
Intervention Acceptability | Through study completion, 6-weeks
  Overall satisfaction with the study

SECONDARY OUTCOMES:
Secondary outcome 1: Knowledge related to dietary sodium | At baseline and at 6-weeks
  To describe the knowledge related to dietary sodium in South Asian Canadians using KAB survey
Secondary outcome 2: Attitudes related to dietary sodium | At baseline and at 6-weeks
  To describe attitudes related to dietary sodium in South Asian Canadians using KAB survey
Secondary outcome 3: Behaviours related to dietary sodium | At baseline and at 6-weeks
  To describe behaviours related to dietary sodium in South Asian Canadians using KAB survey

OTHER OUTCOMES:
Exploratory outcomes-1 | At baseline and at completion of the study-6 weeks
  Systolic BP
Exploratory outcomes-2 | At baseline and at completion of the study-6 weeks
  Diastolic BP
Exploratory outcomes-3 | At baseline and at completion of the study-6 weeks
  24-hour urinary sodium

CONTACTS AND LOCATIONS:
Overall Officials: Salima Hemani, RN, PhD C., Principal Investigator — University of Toronto, Lawrence S. Bloomberg Faculty of Nursing
Locations (1):
- Social Services Network, Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All data will be completely confidential and will not be shared with other researchers.